CLINICAL TRIAL: NCT03750019
Title: Remembered Meal Satisfaction, Satiety and Later Snack Food Intake: A Laboratory Study
Brief Title: Remembered Meal Satisfaction, Satiety and Later Snack Food Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Eric Robinson, Principle Investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RETH000955
Record Dates: First submitted 2018-11-14; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Overweight and Obesity
Keywords: food intake; memory; remembered satisfaction; memory for recent eating; satiety; eating behavior
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Satisfying rehearsal (Experimental): Participants completed the satisfying rehearsal task where they rehearsed the satisfying aspects of the lunchtime meal.
  Interventions: Behavioral: Satisfying rehearsal task
- Dissatisfying rehearsal (Experimental): Participants completed the dissatisfying rehearsal task where they rehearsed the dissatisfying aspects of the lunchtime meal.
  Interventions: Behavioral: Dissatisfying rehearsal task
- Neutral rehearsal (Active Comparator): Participants completed the neutral rehearsal task where they rehearsed their journey to campus that day.
  Interventions: Behavioral: Neutral rehearsal

INTERVENTIONS:
Behavioral: Satisfying rehearsal task — Participants rehearsed satisfying aspects of the lunchtime meal they just ate.
  Arms: Satisfying rehearsal
Behavioral: Dissatisfying rehearsal task — Participants rehearsed dissatisfying aspects of the lunchtime meal they just ate.
  Arms: Dissatisfying rehearsal
Behavioral: Neutral rehearsal — Participants rehearsed their journey to campus that day.
  Arms: Neutral rehearsal

SUMMARY:
This study examined whether remembered meal satisfaction (encompassing memory for meal liking and satiety) can be manipulated in the laboratory and whether this influences later food intake.

DETAILED DESCRIPTION:
This study examined whether remembered meal satisfaction (encompassing memory for meal liking and satiety) can be manipulated in the laboratory and whether this influences later food intake. In a between-subjects design participants consumed a fixed lunch and then rehearsed the satisfying or dissatisfying aspects of the meal, or a neutral experience (control), in order to manipulate memory for meal satisfaction. Three hours later, in a second visit to the laboratory, participants completed a bogus taste-test to measure food intake and meal memory measures.

ELIGIBILITY:
Inclusion Criteria:

* Fluent English
* Not taking medication that affects appetite
* No known history of food allergies or disordered eating

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Ad libitum snack intake | Measured during second visit that took place 3 hours after the baseline visit
  Energy intake (kcal) measured from a bogus taste-test task. Lower intake in those in the satisfying rehearsal condition compared to the control condition and greater intake in the dissatisfying rehearsal condition compared to the control condition were expected.

SECONDARY OUTCOMES:
Memory for general satisfaction | Measured during second visit that took place 3 hours after the baseline visit
  Memory for general satisfaction with the lunchtime meal was measured via five questions: 'Overall, how satisfying did you find the lunchtime meal?', 'Overall, how dissatisfying did you find the lunchtime meal?', 'I liked the lunchtime meal', 'How satisfied were you with the taste of the lunchtime meal?' and 'How dissatisfied were you with the taste of the lunchtime meal?'. Responses were measured using 100-point visual analogue scales with anchors 'not at all' and 'extremely' (0-100). A higher score in those in the satisfying rehearsal condition compared to the control condition and a lower score in the dissatisfying rehearsal condition compared to the control condition were expected.
Memory for satisfaction with meal satiety | Measured during second visit that took place 3 hours after the baseline visit
  Memory for general satisfaction with the lunchtime meal was measured via two questions: 'How satisfied were you with how filling the lunchtime meal was?' and 'How dissatisfied were you with how filling the lunchtime meal was?'. Responses were measured using 100-point visual analogue scales with anchors 'not at all' and 'extremely' (0-100). A higher score in those in the satisfying rehearsal condition compared to the control condition and a lower score in the dissatisfying rehearsal condition compared to the control condition were expected.

OTHER OUTCOMES:
Hunger before lunch | Measured before lunch (during baseline visit)
  Hunger before lunch was measured via a single question asking 'How hungry do you feel right now?'. Responses were measured via a 100-point visual analogue scale with anchors 'not at all' and 'extremely'. No directional hypothesis was made for this outcome.
Hunger after lunch | Measured after lunch (during baseline visit)
  Hunger before lunch was measured via a single question asking 'How hungry do you feel right now?'. Responses were measured via a 100-point visual analogue scale with anchors 'not at all' and 'extremely'. No directional hypothesis was made for this outcome.
Hunger before the bogus taste-test | Measured before the bogus taste-test (in second visit that took place 3 hours after the baseline visit)
  Hunger before lunch was measured via a single question asking 'How hungry do you feel right now?'. Responses were measured via a 100-point visual analogue scale with anchors 'not at all' and 'extremely'. No directional hypothesis was made for this outcome.
Hunger after the bogus taste-test | Measured after the bogus taste-test (in second visit that took place 3 hours after the baseline visit)
  Hunger before lunch was measured via a single question asking 'How hungry do you feel right now?'. Responses were measured via a 100-point visual analogue scale with anchors 'not at all' and 'extremely'. No directional hypothesis was made for this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Robinson, PhD, Principal Investigator — University of Liverpool
Locations (1):
- University of Liverpool, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD is available on the UK Data Service and the study protocol is available on the Open Science Framework.
Supporting Information: Study Protocol
Time Frame: Data is already available.
Access Criteria: There are no restrictions on access to the IPD or study protocol.
URL: http://dx.doi.org/10.5255/UKDA-SN-853370

REFERENCES:
- Available data/document: Individual Participant Data Set: 10.5255/UKDA-SN-853370 — http://dx.doi.org/10.5255/UKDA-SN-853370
- Available data/document: Study Protocol: 10.17605/OSF.IO/WYCKJ — https://doi.org/10.17605/OSF.IO/WYCKJ